CLINICAL TRIAL: NCT03568981
Title: Impact of 5-fraction Stereotactic Partial Breast Irradiation and Whole Breast Irradiation on Cosmetic Outcome and Patient-reported Outcomes in Early-stage Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0160
Record Dates: First submitted 2018-05-15; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Partial Breast Irradiation (PBI): Patients receiving 5-fraction stereotactic partial breast irradiation for breast cancer
  Interventions: Radiation: Partial breast irradiation
- Whole Breast Irradiation (WBI): Patients receiving whole breast irradiation for breast cancer
  Interventions: Radiation: Whole breast irradiation

INTERVENTIONS:
Radiation: Partial breast irradiation — After breast- conservating surgery, all patients are allowed to receive partial breast irradiation or whole breast irradiation after surgery according to the international guidelines and physician's discretion.
  Groups: Partial Breast Irradiation (PBI)
Radiation: Whole breast irradiation — After breast- conservating surgery, all patients are allowed to receive partial breast irradiation or whole breast irradiation after surgery according to the international guidelines and physician's discretion.
  Groups: Whole Breast Irradiation (WBI)

SUMMARY:
This study aim to investigate the effect of 5-fraction stereotactic partial breast irradiation and whole breast irradiation on patient-reported outcomes, cosmetic outcome, and breast tissue fibrosis in early-stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast carcinoma or ductal carcinoma in situ (DCIS)
* Women who underwent breast-conservating surgery and have a plan to undergoing partial or whole breast irradiation
* Good performance status (ECOG 0-1)

Exclusion Criteria:

* Recurrent breast cancer
* History of ipsilateral breast irradiation
* Positive resection margin status after breast surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing radiotherapy after breast-conservating surgery at an academic center
Study Population: Women undergoing radiotherapy after breast-conservating surgery at an academic center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-04-11 (Estimated); Study Completion 2023-04-11 (Estimated)

PRIMARY OUTCOMES:
Change of patient reported psychosocial functioning score | Before radiotherapy (allowed to 8 weeks before radiotherapy)
  Patient reported psychosocial functioning measured in 7 point Likert scale
Change of patient reported psychosocial functioning score | 2 year after radiotherapy (allowed to plus 8 weeks)
  Patient reported psychosocial functioning measured in 7 point Likert scale
Change of patient reported patient treatment satisfaction score | Before radiotherapy (allowed to 8 weeks before radiotherapy)
  Patient reported patient treatment satisfaction measured in 7 point Likert scale
Change of patient reported patient treatment satisfaction score | 2 year after radiotherapy (allowed to plus 8 weeks)
  Patient reported patient treatment satisfaction measured in 7 point Likert scale
Change of patient reported physical functioning score | Before radiotherapy (allowed to 8 weeks before radiotherapy)
  Patient reported physical functioning measured in 7 point Likert scale
Change of patient reported physical functioning score | 2 year after radiotherapy (allowed to plus 8 weeks)
  Patient reported physical functioning measured in 7 point Likert scale
Change of patient reported body image score | Before radiotherapy (allowed to 8 weeks before radiotherapy)
  Patient reported body image score measured in 7 point Likert scale
Change of patient reported body image score | 2 year after radiotherapy (allowed to plus 8 weeks)
  Patient reported body image score measured in 7 point Likert scale
Change of breast cosmesis measures (excellent/good/poor) | Before radiotherapy (allowed to 8 weeks before radiotherapy
  breast cosmesis result is measures by BCCT.core (Breast Cancer Conservative Treatment cosmetic results) software
  - Investigators will whether there are any changes on patient-reported outcomes, cosmetic outcome, and breast tissue fibrosis after radiotherapy. Any differences of theses parameters according to the radiotherapy techniques (PBI vs. WBI) will be examed.
Change of breast cosmesis measures (excellent/good/poor) | 2 year after radiotherapy (allowed to plus 8 weeks)
  breast cosmesis result is measures by BCCT.core (Breast Cancer Conservative Treatment cosmetic results) software
Change of breast-tissue fibrosis measures (gram) | Before radiotherapy (allowed to 8 weeks before radiotherapy
  breast-tissue fibrosis is measured by tissue compliance meter device.
Change of breast-tissue fibrosis measures (gram) | 2 year after radiotherapy (allowed to plus 8 weeks)
  breast-tissue fibrosis is measured by tissue compliance meter device.

SECONDARY OUTCOMES:
Incidence of Radiotherapy-related complications | Before radiotherapy (allowed to 8 weeks before radiotherapy)
  Investigators will check whether there are any kinds of radiotherapy-related complications after PBI or WBI. Any differences of complications according to the radiotherapy techniques will be examed.
Incidence of Radiotherapy-related complications | 2 year after radiotherapy (allowed to plus 8 weeks)
  Investigators will check whether there are any kinds of radiotherapy-related complications after PBI or WBI. Any differences of complications according to the radiotherapy techniques will be examed.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byun HK, Chang JS, Kim H, Kim J, Han MC, Kim SY, Park RH, Kim CJ, Kim YB. Cosmetic Outcome and Toxicity After Stereotactic Accelerated Partial Breast Irradiation in Early Breast Cancer: A Prospective Observational Cohort Study. Int J Radiat Oncol Biol Phys. 2023 Nov 1;117(3):690-700. doi: 10.1016/j.ijrobp.2023.05.018. Epub 2023 May 17. PMID 37201757